CLINICAL TRIAL: NCT03450980
Title: Mobile Medical Application for Cost-effective Strabismus Screening
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Gang Luo, Ph.D., Principal Investigator, Massachusetts Eye and Ear Infirmary
Other Study IDs: 15-061H; 2R44EY025902-02 (NIH)
Record Dates: First submitted 2018-02-07; First posted 2018-03-01 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Strabismus
Keywords: Double Vision, Amblyopia
MeSH Terms: conditions — Strabismus; Diplopia; Amblyopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Strabismus: Participants with strabismus had measurement with the app and compared to the cover test with prism neutralization (gold standard) or eye turning to know eccentricity.

SUMMARY:
Develop and evaluate a new smartphone based app to screen for and measure eye misalignment (strabismus). The investigators will validate the app against simulated strabismus of known magnitude and common clinical tests. They will evaluate the app as a screening tool in high risk populations, to determine the sensitivity and specificity. They hypothesize that the app can measure to within 2 units (prism diopters) of the ground truth, and that it will be correlated with gold standard tests.

DETAILED DESCRIPTION:
The goal of the proposed project is the development and evaluation of a novel mobile medical application for the detection and monitoring of strabismus (eye misalignment). The image analysis technology necessary to measure strabismus using the corneal reflection technique (Photographic Hirschberg Test) has been available for many decades, however it has never been deployed using a smart phone. A smart phone platform will eliminate barriers of cost (since the hardware is maintained and updated by the smart phone industry), leading to rapid wide spread application and allowing the technology to finally reach its potential level of impact for children's eye care in the detection and management of strabismus. Strabismus causes visual confusion and double vision which ultimately results in the brain suppressing vision from the deviated eye. In children this results in under-development (amblyopia) with permanent vision loss in the deviated eye if not detected and treated at a young age. Strabismus in children is also associated with coordination problems such as postural instability and severe social disadvantages. Strabismus develops in an estimated 3-8% of children in the U.S. The prototype smart phone app (Referred to here as the Mobile Eye Alignment App - MEAA), uses photographic analysis of the corneal reflection (Purkinjie image) generated by the smart phone camera flash. The corneal reflection method uses the displacement of the reflection from the center of the pupil in the deviated eye to calculate the amount of eye misalignment. This measurement technique will be deployed for the proposed project using the hardware of the iPhone, a popular phone with an iOS operating system. Preliminary results suggest the app can measure differences in eye alignment of 1.6° (2.8 prism diopters). If successfully developed, the app has potential to be utilized to advance pediatric strabismus research by facilitating and reducing the cost of collecting enormous amounts of data from the general population and under-served or remote populations for epidemiological studies, and allowing researchers to capture eye alignment data much more frequently than is currently possible. Such a tool could better delineate the natural history of strabismus and perhaps help determine its causes. While devices are available which could make these measurements, the costs are prohibitively high (>$3,000 ea.) and will not reach the widespread availability of smart phones. Clinical goals for the app are to provide eye doctors with an objective measurement tool in the exam room, allow daily monitoring of treatment effects, and eventually to be used as a screening tool by school nurses, pediatricians, and parents. The barriers to market success of stand-alone devices is not the accuracy sensitivity or specificity of photographic analysis technique which has been reported with sensitivity from 53% to near 90% and specificity ranging from 76% to 94% for strabismus detection. Impact of strabismus screening for the young - Early detection for strabismus in young children, especially during the critical period up to 2 years of age, is important to ensure that treatment is administered as soon as possible. The success of amblyopia treatment depends on several factors, but principally on the age of onset and the age at which the treatment is initiated. Therapy for amblyopia is maximally effective if started before age 3 and can be initiated as early as 8 months, underscoring the critical need for early and widespread access to strabismus screening. Indeed, countries with long-standing early vision screening programs have reported significantly reduced rates of amblyopia. Access to strabismus screening is also important for older, school age children (age 7-17) suffering from amblyopia, for whom treatment can lead to significant improvements in visual acuity ranging from 20%-70% of patients, depending on their age bracket.

Aims

AIM 1:

Develop and test key functionality of the strabismus app by comparing measurements with successive versions of the prototype app to known angles of eye deviation (non-strabismic volunteers will gaze at off axis targets of known eccentricity).

AIM 2:

Evaluate the strabismus app accuracy and feasibility in participants with strabismus tested with both the app and clinical methods and analyzed for levels of agreement.

Primary Hypothesis: For strabismus ranging from 1 to 30 prism diopters (target range), the optimized version of the app will provide measurements which are highly correlated with the ground truth (simulated strabismus) or clinical tests of eye alignment.

ELIGIBILITY:
Inclusion Criteria:

Ground Truth Aim Study:

* Age 18 to 88 years
* Normal or corrected to normal vision

Clinical Aim Study:

* Ages 18 to 88
* Strabismus
* Able to keep looking at a visual target for 30-60 seconds

Exclusion Criteria:

Ground Truth Aim Study:

* Age less than 18 years or greater than 88.

Clinical Study:

* Age less than 18 or greater than 88
* Inability to keep looking at a visual target for 30-60 seconds

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal vision participants with simulated strabismus and participants with strabismus.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Luo, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Ophthalmology of Clinical Research Office, Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodie SE. Photographic calibration of the Hirschberg test. Invest Ophthalmol Vis Sci. 1987 Apr;28(4):736-42. PMID 3557878
- [Background] Rowe, F.J., Clinical Orthoptics. 3rd ed. 2012: Wiley and Sons. 486.
- [Background] Taylor K, Elliott S. Interventions for strabismic amblyopia. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD006461. doi: 10.1002/14651858.CD006461.pub3. PMID 21833955
- [Background] Cotter SA, Tarczy-Hornoch K, Song E, Lin J, Borchert M, Azen SP, Varma R; Multi-Ethnic Pediatric Eye Disease Study Group. Fixation preference and visual acuity testing in a population-based cohort of preschool children with amblyopia risk factors. Ophthalmology. 2009 Jan;116(1):145-53. doi: 10.1016/j.ophtha.2008.08.031. Epub 2008 Oct 29. PMID 18962921
- [Background] Loudon SE, Rook CA, Nassif DS, Piskun NV, Hunter DG. Rapid, high-accuracy detection of strabismus and amblyopia using the pediatric vision scanner. Invest Ophthalmol Vis Sci. 2011 Jul 7;52(8):5043-8. doi: 10.1167/iovs.11-7503. PMID 21642624
- [Background] Barnard, S. and E. Johnson, Detecting strabismus. Optician, 2013.
- [Background] Klaver P, Marcar V, Martin E. Neurodevelopment of the visual system in typically developing children. Prog Brain Res. 2011;189:113-36. doi: 10.1016/B978-0-444-53884-0.00021-X. PMID 21489386
- [Background] Williams C, Northstone K, Harrad RA, Sparrow JM, Harvey I; ALSPAC Study Team. Amblyopia treatment outcomes after screening before or at age 3 years: follow up from randomised trial. BMJ. 2002 Jun 29;324(7353):1549. doi: 10.1136/bmj.324.7353.1549. PMID 12089090
- [Background] Epelbaum M, Milleret C, Buisseret P, Dufier JL. The sensitive period for strabismic amblyopia in humans. Ophthalmology. 1993 Mar;100(3):323-7. doi: 10.1016/s0161-6420(13)32170-8. PMID 8460000
- [Background] Eibschitz-Tsimhoni M, Friedman T, Naor J, Eibschitz N, Friedman Z. Early screening for amblyogenic risk factors lowers the prevalence and severity of amblyopia. J AAPOS. 2000 Aug;4(4):194-9. doi: 10.1067/mpa.2000.105274. PMID 10951293
- [Background] Lions C, Bui-Quoc E, Bucci MP. Postural control in strabismic children versus non strabismic age-matched children. Graefes Arch Clin Exp Ophthalmol. 2013 Sep;251(9):2219-25. doi: 10.1007/s00417-013-2372-x. Epub 2013 May 9. PMID 23657730
- [Result] Scheiman MM, Hertle RW, Beck RW, Edwards AR, Birch E, Cotter SA, Crouch ER Jr, Cruz OA, Davitt BV, Donahue S, Holmes JM, Lyon DW, Repka MX, Sala NA, Silbert DI, Suh DW, Tamkins SM; Pediatric Eye Disease Investigator Group. Randomized trial of treatment of amblyopia in children aged 7 to 17 years. Arch Ophthalmol. 2005 Apr;123(4):437-47. doi: 10.1001/archopht.123.4.437. PMID 15824215
- [Result] Hertle RW, Scheiman MM, Beck RW, Chandler DL, Bacal DA, Birch E, Chu RH, Holmes JM, Klimek DL, Lee KA, Repka MX, Weakley DR Jr; Pediatric Eye Disease Investigator Group. Stability of visual acuity improvement following discontinuation of amblyopia treatment in children aged 7 to 12 years. Arch Ophthalmol. 2007 May;125(5):655-9. doi: 10.1001/archopht.125.5.655. PMID 17502505
- [Result] Lukman H, Kiat JE, Ganesan A, Chua WL, Khor KL, Choong YF. Negative social reaction to strabismus in school children ages 8-12 years. J AAPOS. 2011 Jun;15(3):238-40. doi: 10.1016/j.jaapos.2011.01.158. Epub 2011 Jun 16. PMID 21683635

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant event.
Groups:
- Participants With Varied Ocular Deviation: This is an observation study, not an intervention study. This was only one group of participants, who were tested for ocular deviation by two methods.. All participants will have eye deviation due to strabismus or gaze shift.
Period: Overall Study
Arm/Group | Participants With Varied Ocular Deviation
Started | 91
Completed | 91
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Normal vision participants with simulated strabismus and participants with strabismus
Groups:
- Participants With Varied Ocular Deviation: This is not an intervention study. There was one time observation using two different tests. Participants with ocular deviation due to either strabismus or gaze shift.
Arm/Group | Participants With Varied Ocular Deviation
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 55
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Undisclosed | 25
  Male | 36
  Female | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comparison of App-measured Eye Deviation Angles to Gold Standard
Description: Linear regression analysis was used to compare the app measurements of strabismus angle to ground truth and gold standard measures. The outcome measure is the difference between the two methods, in terms of least square mean (LSM).
Time Frame: 15 minutes
Population: Participants with Simulated Strabismus and Strabismus
Measure: Least Squares Mean (Standard Deviation); unit: prism diopter
Groups:
- Participants With Ocular Deviation: Participants with eye deviation due to strabismus or gaze shift.
Arm/Group | Participants With Ocular Deviation
Number analyzed (Participants) | 91
prism diopter | 3.3 (4.2)

ADVERSE EVENTS:
Time Frame: Monitored during one study visit, which was typically one hour.
Description: Number of participants at risk is equal to the number enrolled.
Groups:
- Participants With Ocular Deviation: Participants will have eye deviation due to strabismus or gaze shift. There was only one group of participants who were tested by two different methods (prism and app).
Arm/Group | Participants With Ocular Deviation
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03450980/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03450980/SAP_001.pdf